CLINICAL TRIAL: NCT02967640
Title: Does Subacromial Injection With Glutamate Receptor (NMDAR) Antagonist, Ketamine, Attenuate Pain in Rotator Cuff Tendinopathy?
Brief Title: Does Subacromial Injection With Glutamate Receptor Antagonist, Ketamine, Attenuate Pain in Rotator Cuff Tendinopathy?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/1199; 2012-002782-35 (EudraCT Number)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2023-12

CONDITIONS: Rotator Cuff Tendinitis; Chronic Pain
Keywords: Ketamine; Analgesics; Excitatory Amino Acid Antagonists; Receptors, Glutamate; Shoulder
MeSH Terms: conditions — Rotator Cuff Injuries; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketalar (Experimental): ketalar injection, subacromial
  Interventions: Drug: Ketalar; Drug: NaCl 9%
- Placebo (Placebo Comparator): physiological sodium chloride (NaCl 9%) injection, subacromial
  Interventions: Drug: Ketalar; Drug: NaCl 9%

INTERVENTIONS:
Drug: Ketalar — 2,5 ml - if well tolerated immediately followed by another 2,5 ml - of an approximately 1 mg/ml ketalar solution (1 ml of ketalar 10 mg/ml + 9 ml of NaCl 9%) injected 2 times with 1-12 weeks between each injection
  Other Names: Ketamine; Ketanest; Ketaset; Calipsol; Kalipsol; Calypsol
Drug: NaCl 9% — 2,5 ml - if well tolerated immediately followed by another 2,5 ml - of a 9% NaCl solution injected 2 times with 1-12 weeks between each injection

SUMMARY:
The hypothesis of the present study is that in patients with rotator cuff tendinopathy a specific pharmacological blocking of peripheral glutamate-receptor N-methyl-d-aspartate receptor type1 (NMDAR) glutamate receptors will result in pain alleviation. Activated NMDAR1 has been demonstrated to be crucial for pain regulation in various pain disorders, and in biopsies from patients with tendinopathy, NMDAR1 was found to be activated.

To test this hypothesis a specific NMDA receptor antagonist, ketalar (ketamine), will be injected guided by ultrasound into the subacromial space in patients with rotator cuff tendinopathy, and subsequently the pain response will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rotator cuff tendinopathy by exercise-related shoulder pain with positive impingement tests as described by Hawkins and Neers, and MRI findings consistent with tendinopathy.
* Symptom duration at least 1 year to ensure neuronal ingrowth and NMDAR expression

Exclusion Criteria:

* previous surgery in any shoulder.
* previous cortisone use, either as injections or orally
* symptoms or signs of cervicobrachialgia or polyneuropathy
* full thickness rotator cuff ruptures verified by MRI
* primary inflammatory mediated pain, hence, patients with glenohumeral arthrosis, glenohumeral arthritis or systemic disorders predisposing for arthritis
* a central component of pain perception manifested by radiating pain in the involved limb; implying worse outcome after subacromial decompression.
* pregnancy
* breastfeeding
* reduced liver function (Increased serum bilirubin, ASAT or ALAT), decompensated heart failure (NYHA class 3-4)
* increased intracranial pressure or disease of the central nervous system (CNS)
* chronic alcoholism
* epilepsy
* psychiatric disease, increased intraocular pressure
* acute intermittent porphyria
* hyperthyroidism
* use of thyroid hormones
* upper respiratory tract infections
* pneumonia
* intracranial lesions
* acute head injuries
* ocular injuries
* hydrocephalus
* risk factors predisposing for intra-articular bleeding
* increased risk of infection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pain | 30 minutes
  Comparison of pain assessed by a visual analogue scale both at rest and abduction, after selective N-methyl-d-aspartate receptor type 1 blocking by ketalar injection subacromially controlled against Ringer acetate injection.

SECONDARY OUTCOMES:
Pressure pain tolerance | 30 minutes
  Comparison of pressure pain tolerance measured in Lbs/cm3, both at rest and abduction, after selective N-methyl-d-aspartate receptor type 1 blocking by ketalar injection subacromially controlled against Ringer acetate injection.
Supraspinatus pressure pain threshold | 30 minutes
  Comparison of supraspinatus pressure pain threshold measured in Lbs/cm3, after selective N-methyl-d-aspartate receptor type 1 blocking by ketalar injection subacromially controlled against ringer acetate injection

CONTACTS AND LOCATIONS:
Overall Officials: Oystein B Lian, md phd, Study Chair — Helse Nord-Trøndelag HF
Locations (1):
- Department of Orthopedic Surgery, Kristiansund Hospital, Kristiansund, Norway

IPD SHARING:
Plan to Share IPD: No